CLINICAL TRIAL: NCT04168996
Title: Effectiveness of an Individualized Discharge Planning on, Functionality and Quality of Life in Different Severity Rib Fracture Patients
Brief Title: Individualized Discharge Planning in Patients With Rib Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0086UG
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rib fracture patients group (Experimental): Individualized discharge planning in rib fracture patients with different severity of lung injury
  Interventions: Behavioral: Individualized discharge planning
- Control group (No Intervention): Patients included in control group received standard conservative treatment during hospitalization

INTERVENTIONS:
Behavioral: Individualized discharge planning — Discharge planning is designed to ensure healthcare continuity, avoid preventable poor outcomes among at-risk populations, and promote the safe and timely transfer of patient care. The individualized discharge planning is characterized to take into account the preferences, interests and clinical profile of each patient.
  Arms: rib fracture patients group

SUMMARY:
Patients with rib fractures may develop pneumonia and even respiratory failure requiring critical care, ventilator management, and hospitalization. Discharge planning is a broad range of time-limited services designed to ensure healthcare continuity, avoid preventable poor outcomes among at-risk populations, and promote the safe and timely transfer of patients care.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were to be patients hospitalized due to fractures ribs due to falls, traffic accidents, and aggression.

Exclusion Criteria:

* Exclusion criteria were an inability to provide informed consent, the presence of psychiatric or cognitive disorders, progressive neurological disorders, or inability to cooperate. Patients who had experienced hospitalization in the Intense Care Unit were also excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Lung Injury Score (LIS). | Change during the hospitalization, after a week, and after 6 months follow up
  This score was assessed the progression of the lung injury and the development of acute respiratory distress syndrome. The final value was obtained by dividing the sum of the variables used: no injury (LIS=0), mild to moderate (LIS≥0.1), severe (LIS>2.5). We were allocated with a cutoff in the score of LIS.
EuroQol-5D (EQ-5D) | Change during the hospitalization, after a week, and after 6 months follow up
  This measure contains two sections, a descriptive questionnaire about health impairment and a numerical scale about health status perception. The descriptive section includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is categorized into three levels of functioning for each of the five dimensions. The numerical scale ranges from 0 (defined as the worst imaginable health state) to 100 (defined as the best imaginable health state
Barthel Index | Change during the hospitalization, after a week, and after 6 months follow up
  The Barthel Index assesses the level of dependence required by patient to perform the activities. The item scores are totaled which may vary from 0 (total dependence) to 100 (fully independent).

SECONDARY OUTCOMES:
Blaylock Risk Assessment Screening Score (BRASS) | Change during the hospitalization, after a week, and after 6 months follow up
  It comprises a 10-item scale with a score between 0 and 40, with a higher score correlating with a greater likelihood of discharge complications and length of stay.
  A score of 0-10 identifies patients at low risk for complications, 11-20 identifies those requiring discharge planning, and scores above 20 indicate patients who require extensive discharge planning.
Early Screen for Discharge Planning (ESDP) | Change during the hospitalization, after a week, and after 6 months follow up
  The question screening tool was composed for several items (age, living status, disability, and self-reported walking limitation). The score was between 0 and 23. A positive score (≥ 10) was found to indicate the need for automatic referral for complex discharge planning
Newcastle Satisfaction with Nursing Scales (NSNS) | Change during the hospitalization, after a week, and after 6 months follow up
  This measure contains two scales, the experiences of nursing care scale (cognitive evaluation), and the satisfaction with nursing care scale (emotional evaluation). Item scores for each of the scales are summed so that the two scale with scores range from 0 (the best care and full satisfaction) to 100 (the worse care and no satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Granados Santiago M, Valenza MC, Prados Roman E, Lopez Lopez L, Munoz Vigueras N, Cabrera Martos I, Cebria I Iranzo MA. Impacts of tailored, rehabilitation nursing care on functional ability and quality of life in hospitalized elderly patients after rib fractures. Clin Rehabil. 2021 Nov;35(11):1544-1554. doi: 10.1177/02692155211022734. Epub 2021 Jun 6. PMID 34092117